CLINICAL TRIAL: NCT05259605
Title: Observational Study for Assessing Treatment and Outcome of Patients With Primary Brain Tumours Diagnosed According to cIMPACT-NOW Recommendations and the 2021 WHO Classification
Brief Title: Observational Study for Assessing Treatment and Outcome of Patients With Primary Brain Tumours Using cIMPACT-NOW and 2021 WHO Classification
Status: Recruiting | Type: Observational
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-2013-BTG
Record Dates: First submitted 2021-11-22; First posted 2022-02-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Glioma; Glioneuronal Tumor; Choroid Plexus Tumor; Pineal Tumors; Germ Cell Tumor; Tumor of the Sellar Region; Diffuse Midline Glioma, H3 K27M-Mutant; Ependymoma; Embryonal Tumor; Pineal Tumor; Hemangiopericytoma; Hemangioblastoma; Melanocytic Tumor of CNS
Keywords: Rare primary brain tumor; 2021 WHO Classification; molecular diagnosis; Gliomas; Choroid plexus tumors; Embryonal tumors; Pineal tumors
MeSH Terms: conditions — Glioma; Choroid Plexus Neoplasms; Pinealoma; Neoplasms, Germ Cell and Embryonal; Ependymoma; Hemangiopericytoma; Hemangioblastoma | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — * Tumour tissue specifically stored for the purpose of this project
  * Residual biological material ("leftovers") and/or derivatives
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- "Molecular" Gliobastomas, IDH-wildtype: No intervention
  Interventions: Other: Observational
- Paediatric-type diffuse low-grade gliomas: No intervention;
- Paediatric-type diffuse high-grade gliomas: No intervention;
  * diffuse midline glioma, H3 K27-altered
  * diffuse hemispheric glioma, H3 G34-mutant
  * diffuse paediatric-type high-grade glioma, H3-wildtype and IDH-wildtype
  * infant-type hemispheric glioma
- Circumscribed astrocytic gliomas: No intervention
- Glioneuronal and neuronal tumours: No intervention
- Ependymal tumours: No intervention
- Choroid plexus tumours: No intervention
- Embryonal tumours: No intervention;
  * medulloblastoma
  * other
- Pineal tumours: No intervention
- Meningiomas with specific driver mutations and/or grade 3: No intervention
- Mesenchymal, non-meningothelial tumours: No intervention; solitary fibrous tumour hemangioblastomaall all others
- Germ cell tumours: No intervention
- Primary brain tumour with BRAF mutation: No intervention
- Primary brain tumour with NTRK fusion: No intervention
- Primary brain tumour with known germline mutation or family history of a primary brain tumour: No intervention
- Astrocytoma, IDH-mutant, CNS WHO grade 4.: No intervention
- Previously poorly or undefined tumour entities.: No intervention

INTERVENTIONS:
Other: Observational — The goal is to determine whether the new 2021 WHO classification, based on cIMPACT-NOW recommendations, results in more homogeneous patient groups than the old 2016 classification. Furthermore, it will help derive provisional guidelines on how patients with these newly defined tumour entities are best treated. These recommendations will be based on the experience of EORTC investigators with chosen treatments and their experience as reported in this data collection report.
  Groups: "Molecular" Gliobastomas, IDH-wildtype

SUMMARY:
Every new classification depends on its prognostic power and on the type of treatment given. With the rapid evolution of diagnostic methods and the advance in new treatments, there is much less reliable information available on how patients with newly defined brain tumour entities should be treated and what to expect from the current treatments.

The goal is to determine whether the new 2021 WHO classification, based on cIMPACT-NOW recommendations, results in more homogeneous patient groups than the old 2016 classification. Furthermore, it will help derive provisional guidelines on how patients with these newly defined tumour entities are best treated. These recommendations will be based on the experience of EORTC investigators with chosen treatments and their experience as reported in this data collection report.

ELIGIBILITY:
* Age ≥ legal age of consent
* Newly diagnosed or recurrent primary brain tumours within one of the 17 cohorts of interest
* Archival tumour tissue from primary tumour available at the site. Representative tissue from first surgery is preferred, but tissue from surgery for recurrence is allowed. Exception: only tissue from first surgery is allowed for Cohort 16.
* Available MRI/CT scans from primary brain tumour at initial diagnosis
* Patient's consent

Deceased patient:

The clinical data and/or biological material and/or CT/MRI/PET images can be accessed and used if at least one of the following three conditions is met:

* The patient agreed beforehand in his/her lifetime to a further use of his/her data and/or biological material and/or CT/MRI/PET images, or,
* There is consent of a relative to use data and/or biological material and/or CT/MRI/PET images of the deceased patient, or,
* There is a reference to a corresponding legal declaration covering the exemption in case of the impossibility or disproportion of getting access to an informed consent (e.g., causing strain on relatives of deceased patients).

Additionally, in all cases the following three points need to be fulfilled:

* No documentation of previous objection of the patient to the (re-)use of their data, biological material, CT/MR/PET images for research purposes
* A notification to an ethics committee for the re-use of these data, biological material and CT/MRI/PET images
* Any other national requirements are fulfilled, if applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with newly diagnosed or recurrent primary brain tumours, notably those considered to be very rare brain tumours or rare subtypes of common brain tumours will be included. Patients diagnosed between 2011 and 2025.
Sampling Method: Non-Probability Sample
Enrollment: 1650 (Estimated)
Dates: Start 2023-03-21 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2038-07-29 (Estimated)

PRIMARY OUTCOMES:
Best overall and objective response | Followed up for 10 years
  Recorded from the date start of an anti-tumor therapy until disease progression or start of a new anti-tumor therapy.
Progression free survival | Followed up for 10 years
  From the date of start of the anti-tumor therapy until the date of first objective progression as determined by the local investigator or the date of patient's death whichever occurs first. Patients will be followed up for 5 years after enrolment.
Overall Survival | Followed up for 10 years
  Calculated from the date of first pathological diagnosis of the brain tumour; Until the date of death from any cause
Patient and Disease Characteristics | At enrolment and updated every 6 months during follow-up, up to 10 years
  Eligibility, demographics, comorbidities, molecular data

SECONDARY OUTCOMES:
Comparison of patient and disease characteristics between 2016 vs 2021 WHO classifications | At enrolment and during follow-up, up to 10 years
Comparison of treatments and outcomes between classifications | From enrolment through follow-up, up to 10 years
Neuroimaging features at diagnosis and progression | At initial diagnosis and at each documented progression, up to 10 years
Generation of reference datasets for future trials | Throughout study duration, up to 10 years

OTHER OUTCOMES:
Molecular profiling of tumour entities | At diagnosis and/or progression, up to 10 years (depending on tissue availability)
Characterization of rare/undefined tumours (Cohort 17) | At diagnosis and during follow-up, up to 10 years
Next Intervention-Free Survival (NIFS) - Cohort 16 only | From start of anti-tumour therapy until next intervention or death, up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Weller, Principal Investigator — EORTC Study Coordinator
Locations (42):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Universitaetsklinikum Wien - AKH unikliniken, Vienna
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - Institut Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Brussel, Brussels
  - C.H.U. Sart-Tilman, Liège
  - AZ Delta - Campus Rumbeke, Roeselare
- France (3):
  - CHU Lyon - Hopital neurologique Pierre Wertheimer, Lyon
  - Hopital de La Timone, Marseille
  - Hopital la Pitie-Salpetriere, Paris
- Germany (8):
  - Knappschaft Krankenhaus Langendreer, Bochum
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum - Essen, Essen
  - University Hospital Frankfurt -Senckenberg Institute of Neurooncology, Frankfurt
  - Universitaetsklinikum Jena, Jena
  - Universitaetsklinikum Leipzig-Klinik fuer Strahlentherapie und Radioonkologie, Leipzig
  - Universitaetsklinikum Regensburg, Regensburg
- Diagnostic & Therapeutic Center of Athens Hygeia Hospital S.A., Athens, Greece
- Italy (7):
  - Ospedale Bellaria-Bologna, Bologna
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Istituto Neurologico Carlo Besta, Milan
  - IRCCS Ospedale San Raffaele, Milan
  - Istituto Oncologico Veneto, Padua
  - IRCCS-Regina Elena National Cancer Center, Roma
  - Ospedale San Giovanni - Dipartimento Neuroscienze, Torino
- Netherlands (3):
  - The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam
  - Leiden University Medical Centre, Leiden
  - Erasmus MC, Rotterdam
- Oslo University Hospital - Radiumhospitalet, Oslo, Norway
- Portugal (2):
  - Centro Hospitalar Universitario Lisboa Norte - Hospital Sta. Maria, Lisbon
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil - EPE, Lisbon
- Spain (5):
  - Institut Catala d'Oncologia - ICO L'Hospitalet - Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Hospital Germans Trias i Pujol (Institut Catala D'Oncologia), Barcelona
  - Hospital Duran i Reynals, L'Hospitalet de Llobregat
- Switzerland (2):
  - Centre Hospitalier Universitaire Vaudois, Lausanne
  - UniversitaetsSpital Zurich - Neurology Clinic, Zurich
- United Kingdom (3):
  - NHS Lothian - The Royal Infirmary Of Edinburgh, Edinburgh
  - Newcastle Hospitals NHS Trust - Freeman Hospital, Northern Centre For Cancer Care, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham